CLINICAL TRIAL: NCT04163757
Title: The Effects of Crocin Supplementation on Metabolic Parameters, Oxidative Stress, AMP- Activated Protein Kinase and Inflammation-promoting Genes Expression in Peripheral Blood Mononuclear Cells in Patients With Type 2 Diabetes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Nutrition and Food Technology Institute (Other)
Collaborators: Vahideh Behrouz (Unknown); Ali Dastkhosh (Unknown)
Responsible Party: Principal Investigator, Dr Azita Hekmatdoost, Principal Investigator, National Nutrition and Food Technology Institute
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 899
Record Dates: First submitted 2019-11-12; First posted 2019-11-15 (Actual); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — crocin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- placebo (Placebo Comparator)
  Interventions: Dietary Supplement: placebo
- crocin (Active Comparator)
  Interventions: Dietary Supplement: crocin

INTERVENTIONS:
Dietary Supplement: crocin — 2 tablets crocin per day
  Arms: crocin
Dietary Supplement: placebo — 2 tablets placebo per day
  Arms: placebo

SUMMARY:
To study the effects of crocin supplement in patients with type 2 diabetes, 50 patients will be randomly allocated to placebo group and 2 tablets of crocin for 12 weeks. At the first and the end of the intervention, lipid profiles, blood pressure, blood sugar, inflammatory and anthropometric factors will be assessed and compared between groups.

ELIGIBILITY:
Inclusion Criteria:

Age of 40 to 65 years type 2 diabetes: and body mass index range of 18.5 to 30 kg/m2

Exclusion Criteria:

pregnancy or lactation A history of Cardiovascular disease, Pulmonary disease, Renal disease

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2019-01-20 (Actual); Primary Completion 2019-03-06 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
type 2 diabetes | 12 weeks
  number of participants with normal plasma glucose

CONTACTS AND LOCATIONS:
Locations (1):
- National Nutrition and Food Technology Research Institute, Tehran, Iran

REFERENCES:
- [Derived] Behrouz V, Dastkhosh A, Hedayati M, Sedaghat M, Sharafkhah M, Sohrab G. The effect of crocin supplementation on glycemic control, insulin resistance and active AMPK levels in patients with type 2 diabetes: a pilot study. Diabetol Metab Syndr. 2020 Jul 9;12:59. doi: 10.1186/s13098-020-00568-6. eCollection 2020. PMID 32670418